CLINICAL TRIAL: NCT00380276
Title: Open Label Study of the Effect of Daily Treatment With MPC-7869 in Subjects With Dementia of the Alzheimer's Type
Brief Title: Open-Label Treatment With MPC-7869 for Patients With Alzheimer's Who Previously Participated in an MPC-7869 Protocol
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Myriad has discontinued the development of Flurizan.
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Ed Swabb, MD, Myriad Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-7869-05-009
Record Dates: First submitted 2006-09-21; First posted 2006-09-25 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; Dementia; Dementia of Alzheimer Type
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — tarenflurbil

ARMS (1):
- Open Label Arm (Other): Treatment is open-label
  Interventions: Drug: MPC-7869

INTERVENTIONS:
Drug: MPC-7869 — 800 mg BID Oral dosing

SUMMARY:
Open-label treatment with MPC-7869 for participants in a previous randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a previous MPC-7869 randomized protocol
* Have had a diagnosis of probable Alzheimer's disease.
* Men or women ages 55 years or greater and living in the community at the time of enrollment (i.e., not living in a rest home or nursing care facility).
* Signed the subject Informed Consent Form and is willing and able to participate for the duration of the study.
* Female subjects must be surgically sterile or postmenopausal for > 1 year.
* Subjects must have a reliable caregiver who can read, understand and speak English or Spanish.

Exclusion Criteria:

* History or evidence of, active malignancy, except for basal cell carcinoma or squamous cell carcinoma of the skin, within the 24 months prior to entry. Men with prostate cancer may be enrolled at the discretion of the sponsor.
* Chronic or acute renal, hepatic or metabolic disorder.
* Use of any investigational therapy within 30 days, or 5 half-lives, whichever is longer, and/or use of AD immunotherapy prior to screening.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety | For study duration

CONTACTS AND LOCATIONS:
Overall Officials: Mark Laughlin, MD, Study Director — Myrexis Inc.
Locations (90):
- United States (84):
  - Alabaster, Alabama
  - Huntsville, Alabama
  - Phoenix, Arizona
  - Sun City, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - Irvine, California
  - Lafayette, California
  - Laguna Hills, California
  - Long Beach, California
  - Rancho Mirage, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Vista, California
  - Danbury, Connecticut
  - Darien, Connecticut
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Deerfield Beach, Florida
  - Fort Meyers, Florida
  - Fort Myers, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Naples, Florida
  - Sunrise, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - West Yarmouth, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Rochester, Minnesota
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Kenilworth, New Jersey
  - Morristown, New Jersey
  - Princeton, New Jersey
  - Stratford, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Brooklyn, New York
  - Elmsford, New York
  - New York, New York
  - Olean, New York
  - Rochester, New York
  - Syracuse, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Centerville, Ohio
  - Columbus, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Jenkintown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Scotland, Pennsylvania
  - East Providence, Rhode Island
  - Beaufort, South Carolina
  - Charleston, South Carolina
  - Greer, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Alexandria, Virginia
  - Charlottesville, Virginia
  - Virginia Beach, Virginia
  - Middleton, Wisconsin
  - Milwaukee, Wisconsin
- Canada (6):
  - Winnepeg, Manitoba
  - Halifax, Nova Scotia
  - Kingston, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Regina, Saskatchewan